CLINICAL TRIAL: NCT03420443
Title: Randomized Clinical Trial of Effects of Synbiotics on Intestinal Microbiota in Patients Undergoing Short-course Preoperative Radiotherapy During Treatment of Rectal Cancer
Brief Title: Action of Synbiotics on Irradiated GI Mucosa in Rectal Cancer Treatment
Acronym: FIPIREX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: LU1007-3
Record Dates: First submitted 2017-11-08; First posted 2018-02-05 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Rectal Cancer
Keywords: radiotherapy, probiotics
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Oat bran (Experimental): 45 g oat bran
  Interventions: Dietary Supplement: Oat bran
- Oat bran and blueberry husks (Experimental): 13 g freeze dried blueberry husks and 22 g oat bran + probiotic bacteria.
  Interventions: Dietary Supplement: Oat bran and blueberry husks
- No oral supplementation (Other): No oral supplementation.
  Interventions: Dietary Supplement: No oral supplementation

INTERVENTIONS:
Dietary Supplement: Oat bran — 45 g oat bran.
  Arms: Oat bran
Dietary Supplement: Oat bran and blueberry husks — 13 g freeze dried blueberry husks and 22 g oat bra + probiotic bacteria.
  Arms: Oat bran and blueberry husks
Dietary Supplement: No oral supplementation — No oral supplementation.
  Arms: No oral supplementation

SUMMARY:
The aim of this study is to investigate how bacteria and fibre interact with the epithelial cells of the gastrointestinal mucosa to reduce inflammation and to diminish tissue damage caused by radiation therapy to patients diagnosed with rectal cancer.

DETAILED DESCRIPTION:
Thirty patients diagnosed with rectal cancer receiving short term radiation therapy 25 Gray (Gy) during one week preoperatively will be examined. The patients will be divided into three groups with ten patients in each group. One control group without no treatment/study product, one group receiving a test product of 45 g of oat bran and freezing medium only, and one group having a probiotic bacteria, Lactobacillus plantarum HEAL 19 (1010 CFU/g), freezed dried blueberry husks (13 g) and oat bran (22 g), corresponding to 8 g fibre per day in each of the two treated groups. The patients will consume the test product once a day 1 week before and during radiotherapy (2 weeks in total). Mucosal biopsies for microflora analysis and blood samples for analysis of SCFAs and cytokines will be collected at inclusion as well as faecal samples. After radiation therapy, at surgery, blood samples, faecal samples and mucosal biopsies are collected. Fresh faecal samples, blood samples and mucosal biopsies are stored at -80°C until analysis.

ELIGIBILITY:
Inclusion Criteria:

* Rectal cancer/Adenocarcinoma recti
* Informed Consent explained orally and written, understood, agreed and signed

Exclusion Criteria:

* Diabetes Mellitus
* Inflammatory bowel disease
* Previous radiation to pelvis area
* Ongoing steroid or immunosuppressive therapy
* Ongoing antibiotics therapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-11; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Action of synbiotics on irradiated GI mucosa in rectal cancer treatment | 2 weeks
  Reaction of gastrointestinal mucosa in a clinical setting in patients with preoperative radiotherapy treatment of rectal cancer pre-treated with either a probiotic bacteria, blueberry husks and oat bran, oat bran only or no pre-treatment at all, measured by analysis of bacterial diversity.
Action of synbiotics on irradiated GI mucosa in rectal cancer treatment | 2 weeks
  Reaction of gastrointestinal mucosa in a clinical setting in patients with preoperative radiotherapy treatment of rectal cancer pre-treated with either a probiotic bacteria, blueberry husks and oat bran, oat bran only or no pre-treatment at all, measured by analysis of inflammation.

CONTACTS AND LOCATIONS:
Overall Officials: Bengt Jeppsson, Prof, Principal Investigator — University of Lund, Sweden

IPD SHARING:
Plan to Share IPD: No